CLINICAL TRIAL: NCT02306252
Title: LCCC 1409: The CARE Program: CAncer REhabilitation Pilot Study for Older Adults
Brief Title: The CARE Program: CAncer REhabilitation Pilot Study for Older Adults
Acronym: CARE Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LCCC1409; 14-1159 (Other: University of North Carolina IRB)
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Cancer
Keywords: Cancer; Older Adult; Geriatric; Function; Functional Deficit; Occupational Therapy; Physical Therapy; Supportive Care; Oncology; physiology; Geriatric Assessment; Health Services for the Aged; Physical Therapy Specialty
MeSH Terms: conditions — Neoplasms | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CARE Intervention (Experimental): This group will be contacted to make an appointment for outpatient Occupational and Physical therapy. The therapist will determine the type, frequency and length of treatment. Follow up phone calls will be made to ensure appointments are made, kept and rescheduled as needed.
  Interventions: Other: Occupational and Physical Therapy
- CARE Control (No Intervention): Patients randomized to this arm will receive contact information and a brochure outlining the services available within the supportive care program. The study coordinator will provide the information based on their results and assist the patient with contacting the program if desired.

INTERVENTIONS:
Other: Occupational and Physical Therapy — OT and PT will be arranged for the subject and conducted in a manner as determined by the therapist.
  Arms: CARE Intervention

SUMMARY:
The CARE Program is a randomized trial of a cancer rehabilitation program designed to help older cancer patients who have shown to have a loss of function.

DETAILED DESCRIPTION:
This is a prospective, two-arm, single-center randomized controlled pilot trial of a cancer rehabilitation program for older adults, titled the 'CARE program,' which is designed to maintain and/or improve functional status and quality of life in older adults diagnosed with cancer. Adults aged 65 years and older with cancer will be screened with a Geriatric Assessment (GA) for eligibility. Although breast cancer patients will be eligible, this study will focus primarily on other types of cancers. Adults with at least one functional deficit --defined as impairment in ability to perform activities of daily living or instrumental activities of daily living, cognitive decline or balance -- will be randomized to either the intervention (CARE program) or to the control arm (Supportive care services information only). Both arms will receive a brochure about the supportive care program to provide patients who we've identified as having deficits with information about auxiliary services available and because the intent is to limit the difference between the groups. We hypothesize that patients who participate in the CARE program will maintain or improve functional status and quality of life when compared to supportive care services information only.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older
* Has an outpatient appointment within UNC Chapel Hill Lineberger Comprehensive Cancer Center
* Diagnosis of cancer within last two years.
* Has a life expectancy of 12 months or longer. All cancer types are included.
* English speaking
* Willing to complete the UNC GA
* Has at least one functional deficit as defined by GA screen
* Understands study design, risks, and benefits and have signed informed consent
* Willing to be randomized into either study arm
* Ability to safely participate in outpatient rehabilitation program

Exclusion Criteria:

* Unable to safely participate in outpatient rehabilitation.
* Currently receiving rehabilitation.
* Any participant who has urologic cancer or is enrolled in a competing trial.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 67 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
To measure the change in Nottingham Extended Activities of Daily Living (NEADL) score from baseline to three months. | 3 months
  Compare the change in NEADL scores from baseline to 3 months between patients who receive the CARE program (intervention) and those in the control arm.

SECONDARY OUTCOMES:
To measure the change in Activities of Daily Living from Baseline and 2 months | 2 months
  As measured by the Geriatric Assessment
To measure the change in Activities of Daily Living from Baseline and 3 months | 3 months
  As measured by the Geriatric Assessment
To measure the change in physical health from Baseline and 3 months | 3 months
  As measured by the Geriatric Assessment
To measure the change in physical health from Baseline and 2 months | 2 months
  As measured by the Geriatric Assessment
To measure the change in quality of life from Baseline and 2 months | 2 months
  As measured by the PROMIS assessment
To measure the change in quality of life from Baseline and 3 months | 3 months
  As measured by the PROMIS assessment
To measure the change in internalized occupational possibilities from Baseline and 3 months | 3 months
  As measured by the Possibilities for Activity Scale (PActS)
To measure the change in internalized occupational possibilities from Baseline and 2 months | 2 months
  As measured by the Possibilities for Activity Scale (PActS)
To measure the change in cognitive function from Baseline and 2 months | 2 months
  As measured by the Blessed Memory Orientation Concentration test
To measure the change in cognitive function from Baseline and 3 months | 3 months
  As measured by the Blessed Memory Orientation Concentration test
To measure the feasibility of the CARE Program | 3 months
  To describe the feasibility of the CARE program by reporting enrollment and retention as defined by (1) percent eligible who agree to participate (2) percent in each group that completed follow-up measures at 2 and 3 months and (3) percent of patients in CARE program who go to 70% of appointments.
To measure the change in balance over the course of the study | 3 months
  Intervention Group Only: As measured by the Berg Balance Scale
To measure the change in upper extremity use and ability over the course of the study | 3 months
  Intervention Group Only: As measured by the Disability of the Arm, Shoulder and Hand scale
To measure the change in cognition over the course of the study | 3 months
  Intervention Group Only: As measured by the Montreal Cognitive Assessment
To measure the change in dynamic gait ability over the course of the study | 3 months
  Intervention Group Only: As measured by the Dynamic Gait Index
To measure satisfaction with the CARE Program | 3 months
  To evaluate the program a short interview will be completed with CARE team to determine what worked well, what didn't and suggested changes/improvements for CARE program after completion of project.

CONTACTS AND LOCATIONS:
Overall Officials: Mackenzi Pergolotti, PhD, Principal Investigator — Colorado State University
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States